CLINICAL TRIAL: NCT03725202
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of Upadacitinib in Subjects With Giant Cell Arteritis: SELECT-GCA
Brief Title: A Study to Evaluate the Safety and Efficacy of Upadacitinib in Participants With Giant Cell Arteritis
Acronym: SELECT-GCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-852; 2023-505476-29-00 (Other: EU CT); 2017-003978-13 (EudraCT Number)
Record Dates: First submitted 2018-10-27; First posted 2018-10-30 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Giant Cell Arteritis (GCA)
Keywords: Giant Cell Arteritis (GCA); ABT-494; Upadacitinib
MeSH Terms: conditions — Giant Cell Arteritis | interventions — upadacitinib; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Placebo + 52-week CS taper (Placebo Comparator): Participants received placebo tablets for upadacitinib administered orally once daily (QD) for 52 weeks and a 52-week corticosteroid (CS) taper regimen during Period 1.
  Interventions: Drug: Corticosteroid (CS); Other: Placebo
- 7.5 mg Upadacitinib + 26-week CS taper (Experimental): Participants received 7.5 mg upadacitinib tablets administered orally once daily (QD) for 52 weeks and a 26-week corticosteroid (CS) taper regimen during Period 1.
  Interventions: Drug: Upadacitinib; Drug: Corticosteroid (CS)
- 15 mg Upadacitinib + 26-week CS taper (Experimental): Participants received 15 mg upadacitinib tablets administered orally once daily (QD) for 52 weeks and a 26-week corticosteroid (CS) taper regimen during Period 1.
  Interventions: Drug: Upadacitinib; Drug: Corticosteroid (CS)
- Placebo + 52-week CS taper -> Placebo (Placebo Comparator): Participants who achieved sustained remission for at least 24 weeks prior to the Week 52 visit (at the end of Period 1) OR at remission at the Week 52 visit only who were assigned to placebo tablets for upadacitinib administered orally once daily (QD) in Period 1 continued to receive placebo tablets for upadacitinib administered orally once daily (QD) in Period 2.
  Interventions: Other: Placebo
- 7.5 mg Upadacitinib + 26-week CS taper -> 7.5 mg Upadacitinib (Experimental): Participants received 7.5 mg upadacitinib tablets administered orally once daily (QD) in Period 2.
  Interventions: Drug: Upadacitinib
- 7.5 mg Upadacitinib + 26-week CS taper -> Placebo (Experimental): Participants received placebo tablets for upadacitinib administered orally once daily (QD) in Period 2.
  Interventions: Other: Placebo
- 15 mg Upadacitinib + 26-week CS taper -> 15 mg Upadacitinib (Experimental): Participants received 15 mg upadacitinib tablets administered orally once daily (QD) in Period 2.
  Interventions: Drug: Upadacitinib
- 15 mg Upadacitinib + 26-week CS taper -> Placebo (Experimental): Participants received placebo tablets for upadacitinib administered orally once daily (QD) in Period 2.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Upadacitinib — Administered orally once a day
  Other Names: ABT-494; RINVOQ
  Arms: 15 mg Upadacitinib + 26-week CS taper; 15 mg Upadacitinib + 26-week CS taper -> 15 mg Upadacitinib; 7.5 mg Upadacitinib + 26-week CS taper; 7.5 mg Upadacitinib + 26-week CS taper -> 7.5 mg Upadacitinib
Drug: Corticosteroid (CS) — At Baseline, all participants switched to corticosteroids (CS) provided by the sponsor with the oral prednisone or prednisolone dose at 20, 30, 40, 50, or 60 mg QD. The initial dose of prednisone or prednisolone was at the discretion of the investigator, based on disease severity and comorbid medical conditions, at a minimum of 20 mg QD at Baseline. At Baseline, if a participant was on a dose other than 20, 30, 40, 50, or 60 mg QD, the dose was rounded up or down, as clinically indicated per investigator discretion, to the nearest of these doses. Prednisone or prednisolone was tapered according to a predefined schedule over a 26- or 52-week period. Open-label prednisone or prednisolone was provided until the dose was tapered to 20 mg/day. Subsequently, blinded prednisone or prednisolone was provided for the remaining blinded taper regimen through Week 52.
  Arms: 15 mg Upadacitinib + 26-week CS taper; 7.5 mg Upadacitinib + 26-week CS taper; Placebo + 52-week CS taper
Other: Placebo — Administered orally once a day
  Arms: 15 mg Upadacitinib + 26-week CS taper -> Placebo; 7.5 mg Upadacitinib + 26-week CS taper -> Placebo; Placebo + 52-week CS taper; Placebo + 52-week CS taper -> Placebo

SUMMARY:
This study consists of two periods. The objective of Period 1 is to evaluate the efficacy of upadacitinib in combination with a 26-week corticosteroid (CS) taper regimen compared to placebo in combination with a 52-week CS taper regimen, as measured by the proportion of participants in sustained remission at Week 52, and to assess the safety and tolerability of upadacitinib in participants with giant cell arteritis (GCA). The objective of Period 2 is to evaluate the safety and efficacy of continuing versus withdrawing upadacitinib in maintaining remission in participants who achieved sustained remission in Period 1.

Safety and efficacy data through 06 February 2024 are included in the interim analysis, which was conducted after all participants completed the Week 52 visit or discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of giant cell arteritis (GCA) according to the following criteria:

  * History of erythrocyte sedimentation rate (ESR) >= 50 mm/hour or high sensitivity C-reactive protein (hsCRP)/CRP >=1.0 mg/dL
  * Presence of at least one of the following: Unequivocal cranial symptoms of GCA or Unequivocal symptoms of polymyalgia rheumatica (PMR)
  * Presence of at least one of the following: temporal artery biopsy revealing features of GCA or evidence of large vessel vasculitis by angiography or cross-sectional imaging such as ultrasound, magnetic resonance imaging (MRI), computed tomography (CT) or positron emission tomography (PET).
* Active GCA, either new onset or relapsing, within 8 weeks of Baseline.
* Participants must have received treatment with >=40 mg prednisone (or equivalent) at any time prior to Baseline and be receiving prednisone (or equivalent) >= 20 mg once daily (QD) at Baseline.
* Participants must have GCA that, in the opinion of the investigator, is clinically stable to allow the participant to safely initiate the protocol-defined corticosteroid (CS) taper regimen.
* Females must either be postmenopausal or permanently surgically sterile or, practicing at least 1 specified method of birth control through the study.

Exclusion Criteria:

* Prior exposure to any Janus Kinase (JAK) inhibitor.
* Treatment with an interleukin-6 (IL-6) inhibitor within 4 weeks of study start, or prior treatment with an IL-6 inhibitor and experienced a disease flare during treatment.
* Use of any of the following systemic immunosuppressant treatments within the specified timeframe prior to study start:

  * Anakinra within 1 week of study start.
  * Methotrexate, hydroxychloroquine, cyclosporine, azathioprine, or mycophenolate within 4 weeks of study start.
  * Oral corticosteroid (CS) for conditions other than GCA within 4 week of study start, or intravenous CS within 4 weeks of study start.
  * Greater than or equal to 8 weeks for leflunomide if no elimination procedure was followed, or adhere to an elimination procedure.
  * Cell-depleting agents or alkylating agents including cyclophosphamide within 6 months of study start.
* Current or past history of infection including herpes zoster or herpes simplex, human immunodeficiency virus (HIV), active Tuberculosis, active or chronic recurring infection, active hepatitis B or C.
* Female who is pregnant, breastfeeding, or considering pregnancy during the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2025-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (172):
- United States (53):
  - Rheum Assoc of North Alabama /ID# 168668, Huntsville, Alabama
  - Arizona Arthritis and Rheumatology Research - Glendale Office /ID# 204702, Glendale, Arizona
  - VA Long Beach Healthcare System /ID# 203833, Long Beach, California
  - Robin K. Dore MD, Inc /ID# 201950, Tustin, California
  - Denver Arthritis Clinic /ID# 171552, Denver, Colorado
  - Duplicate_Western Connecticut Health Network- Germantown Rd /ID# 205071, Danbury, Connecticut
  - Rheumatology Associates of South Florida (RASF) - Clinical Research /ID# 169040, Boca Raton, Florida
  - Lakes Research, LLC /ID# 210442, Miami, Florida
  - Ctr Arthritis & Rheumatic Dise /ID# 168667, Miami, Florida
  - Medallion Clinical Research Institute, LLC /ID# 168666, Naples, Florida
  - Omega Research Group /ID# 201903, Orlando, Florida
  - IRIS Research and Development, LLC /ID# 169406, Plantation, Florida
  - Clinical Research of West Florida - Tampa /ID# 201899, Tampa, Florida
  - Clinical Research of West Florida, Inc /ID# 201901, Tampa, Florida
  - Duplicate_University of South Florida /ID# 207077, Tampa, Florida
  - Lovelace Scientific Resources /ID# 169041, Venice, Florida
  - Arthritis and Rheumatology /ID# 170295, Atlanta, Georgia
  - Institute of Arthritis Research /ID# 168490, Idaho Falls, Idaho
  - Duplicate_Rush University Medical Center /ID# 224581, Chicago, Illinois
  - Ochsner Clinic Foundation /ID# 200723, Baton Rouge, Louisiana
  - The Arthritis & Diabetes Clinic, Inc. /ID# 171199, Monroe, Louisiana
  - Ochsner Clinic Foundation-New Orleans /ID# 171200, New Orleans, Louisiana
  - Louisiana State Univ HSC /ID# 202646, Shreveport, Louisiana
  - Rheumatology Associates PA - Portland /ID# 225011, Portland, Maine
  - The Center for Rheumatology and Bone Research /ID# 168652, Wheaton, Maryland
  - University of Michigan Hospitals /ID# 168645, Ann Arbor, Michigan
  - Wayne State University Health Center /ID# 212755, Detroit, Michigan
  - Henry Ford Medical Center - New Center One /ID# 207456, Detroit, Michigan
  - Duplicate_AA Medical Research Center - Grand Blanc /ID# 201854, Grand Blanc, Michigan
  - Duplicate_West Michigan Rheumatology /ID# 168647, Grand Rapids, Michigan
  - Clinvest Research LLC /ID# 208182, Springfield, Missouri
  - Physician Research Collaboration, LLC /ID# 168610, Lincoln, Nebraska
  - University Clinical Research Center /ID# 202504, Somerset, New Jersey
  - University of Rochester Medical Center /ID# 213527, Rochester, New York
  - Marietta Memorial Hospital /ID# 210834, Marietta, Ohio
  - STAT Research, Inc. /ID# 200436, Vandalia, Ohio
  - University of Pennsylvania /ID# 168655, Philadelphia, Pennsylvania
  - Piedmont Arthritis Clinic, PA /ID# 212431, Greenville, South Carolina
  - Articularis Healthcare Group, Inc d/b/a Low Country Rheumatology /ID# 212761, Summerville, South Carolina
  - West Tennessee Research Institute /ID# 209256, Jackson, Tennessee
  - Arthritis Associates of Kingsport /ID# 212756, Kingsport, Tennessee
  - Allen Arthritis /ID# 225527, Allen, Texas
  - Tekton Research, L.L.C /ID# 201801, Austin, Texas
  - Precision Comprehensive Clinical Research Solutions /ID# 201798, Colleyville, Texas
  - West Texas Clinical Research /ID# 204834, Lubbock, Texas
  - Arthritis and Rheumatology Institute, PLLC /ID# 214612, Plano, Texas
  - Baylor Scott & White Center for Diagnostic Medicine /ID# 213529, Temple, Texas
  - University of Vermont Medical Center /ID# 211179, Burlington, Vermont
  - Carilion Clinic /ID# 212928, Roanoke, Virginia
  - Kadlec Clinic Rheumatology /ID# 201618, Kennewick, Washington
  - University of Washington /ID# 201619, Seattle, Washington
  - Aurora Rheumatology and Immunotherapy Center /ID# 201853, Franklin, Wisconsin
  - Froedtert Memorial Lutheran Hospital /ID# 224557, Milwaukee, Wisconsin
- Australia (6):
  - Emeritus Research Sydney /ID# 201937, Botany, New South Wales
  - Prince of Wales Hospital /ID# 210995, Randwick, New South Wales
  - Griffith University /ID# 223829, Southport, Queensland
  - The Queen Elizabeth Hospital /ID# 201939, Woodville South, South Australia
  - Emeritus Research /ID# 201938, Camberwell, Victoria
  - Fiona Stanley Hospital /ID# 201941, Murdoch, Western Australia
- Austria (2):
  - Medizinische Universitaet Innsbruck /ID# 201786, Innsbruck, Tyrol
  - Rheuma-Zentrum Wien-Oberlaa GmbH /ID# 201781, Vienna, Vienna
- Belgium (3):
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant /ID# 224334, Yvoir, Namur
  - UZ Gent /ID# 202778, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 202779, Leuven, Vlaams-Brabant
- Canada (5):
  - Duplicate_University of Alberta Hospital - Division of Hematology /ID# 208629, Edmonton, Alberta
  - St. Joseph's Healthcare /ID# 204160, Hamilton, Ontario
  - CISSSBSL -Hopital regional de Rimouski /ID# 224266, Rimouski, Quebec
  - Centre de Recherche Musculo-Squelettique /ID# 201224, Trois-Rivières, Quebec
  - Rheumatology Associates /ID# 201843, Saskatoon, Saskatchewan
- Czechia (3):
  - Fakultni nemocnice Olomouc /ID# 202041, Olomouc
  - Axon Clinical, s.r.o. /ID# 202468, Prague
  - Medical Plus, s.r.o. /ID# 200865, Uherské Hradiště
- Denmark (2):
  - Aarhus University Hospital /ID# 171177, Aarhus C, Central Jutland
  - Sydvestjysk Sygehus /ID# 200216, Esbjerg, Region Syddanmark
- France (11):
  - Hopital Saint Joseph /ID# 171540, Marseille, Bouches-du-Rhone
  - CHU Dijon /ID# 225277, Dijon, Cote-d Or
  - Hopital de la Cavale Blanche /ID# 171549, Brest, Finistere
  - CHU Toulouse - Hopital Purpan /ID# 171547, Toulouse, Haute-Garonne
  - CHRU Lille - Hopital Claude Huriez /ID# 171543, Lille, Nord
  - Hopitaux Universitaires Paris Centre-Hopital Cochin /ID# 171545, Paris, Paris
  - CHU de Nantes, Hotel Dieu -HME /ID# 171544, Nantes, Pays de la Loire Region
  - HCL - Hopital de la Croix-Rousse /ID# 211184, Lyon, Rhone
  - CHU de CAEN - Hopital de la Cote de Nacre /ID# 171539, Caen
  - CHRU Tours - Hopital Trousseau /ID# 245232, Chambray-lès-Tours
  - Hopital Pitie Salpetriere /ID# 171542, Paris, Île-de-France Region
- Germany (6):
  - Medius Klinik Kirchheim /ID# 200637, Kirchheim unter Teck, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen /ID# 223854, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Wuerzburg /ID# 213340, Würzburg, Bavaria
  - Immanuel Krankenhaus Berlin /ID# 223855, Buch
  - Medizinische Versorgungszentren Burghausen Altoetting /ID# 208773, Burghausen
  - Medizinische Hochschule Hannover /ID# 200632, Hanover
- Greece (3):
  - General Hospital of Athens Gennimatas /ID# 210129, Athens, Attica
  - General Hospital of Athens Ippokratio /ID# 202181, Athens, Attica
  - 424 General MILITARY Hospital /ID# 210973, Efkarpia (Thessalonikis), Thessaloniki
- Hungary (4):
  - Debreceni Egyetem-Klinikai Kozpont /ID# 201526, Debrecen, Hajdú-Bihar
  - Betegapolo Irgalmasrend Budai Irgalmasrendi Korhaz /ID# 204018, Budapest
  - Orszagos Reumatologiai es Fizioterapias Intezet /ID# 211454, Budapest
  - Del-Budai Centrumkorhaz Szent Imre Egyetemi Oktatokorhaz /ID# 201838, Budapest
- Israel (3):
  - Bnai Zion Medical Center /ID# 240733, Haifa, H_efa
  - The Lady Davis Carmel Medical Center /ID# 240731, Haifa, H_efa
  - The Chaim Sheba Medical Center /ID# 241041, Ramat Gan, Tel Aviv
- Italy (3):
  - Azienda Sanitaria dell'Alto Adige /ID# 200081, Bolzano
  - Azienda Ospedaliero-Universitaria di Modena /ID# 200079, Modena
  - Azienda Ospedaliera Universitaria Friuli Centrale/Presidio Ospedaliero Universit /ID# 200082, Udine
- Japan (10):
  - Japan Organization of Occupational Health and Safety Chubu Rosai Hospital /ID# 202946, Nagoya, Aichi-ken
  - Kagawa University Hospital /ID# 200171, Kita-gun, Kagawa-ken
  - St. Marianna University Hospital /ID# 218692, Kawasaki-shi, Kanagawa
  - Duplicate_Japanese Red Cross Kumamoto Hospital /ID# 203507, Kumamoto, Kumamoto
  - Tohoku University Hospital /ID# 200172, Sendai, Miyagi
  - Okayama University Hospital /ID# 203156, Okayama, Okayama-ken
  - Tomishiro Central Hospital /ID# 203897, Tomigusuku-shi, Okinawa
  - Sakai City Medical Center /ID# 202643, Sakai-shi, Osaka
  - Duplicate_Jichi Medical University Hosp /ID# 200169, Shimotsuke-shi, Tochigi
  - St.Luke's International Hospital /ID# 200170, Chuo-ku, Tokyo
- Netherlands (6):
  - Radboud Universitair Medisch Centrum /ID# 212925, Nijmegen, Gelderland
  - Zuyderland Medisch Centrum /ID# 224551, Heerlen, Limburg
  - ZiekenhuisGroep Twente /ID# 200038, Almelo, Overijssel
  - Medisch Centrum Leeuwarden /ID# 201716, Leeuwarden, Provincie Friesland
  - Duplicate_Erasmus Medisch Centrum /ID# 201717, Rotterdam, South Holland
  - Universitair Medisch Centrum Groningen /ID# 201715, Groningen
- New Zealand (6):
  - Optimal Clinical Trials Ltd /ID# 201946, Grafotn, Auckland
  - Aotearoa Clinical Trials /ID# 201942, Papatoetoe, Auckland
  - Timaru Medical Specialists Ltd /ID# 201943, Timaru, Canterbury
  - Waikato Hospital /ID# 201944, Hamilton, Waikato Region
  - CGM Research Trust /ID# 224061, Christchurch Central
  - Porter Rheumatology Ltd /ID# 223830, Nelson
- Norway (3):
  - Drammen Sykehus /ID# 201560, Drammen, Buskerud
  - Haukeland universitetssjukehus /ID# 201602, Bergen, Hordaland
  - Rikshospitalet OUS HF /ID# 202004, Oslo
- Portugal (4):
  - Unidade Local de Saude de Gaia/Espinho, EPE /ID# 208151, Vila Nova de Gaia, Porto District
  - Unidade Local de Saúde do Alto Minho, EPE - Hospital Conde de Bertiandos /ID# 205186, Ponte de Lima, Viana do Castelo District
  - Unidade Local de Saúde da Guarda, EPE /ID# 224878, Guarda
  - Unidade Local de Saude de Santa Maria, EPE /ID# 203530, Lisbon
- Romania (4):
  - Spitalul Clinic Judetean de Urgenta Cluj -Napoca /ID# 204887, Cluj-Napoca, Cluj
  - Cabinet Medical Dr. Avram S.R.L /ID# 224336, Timișoara, Timiș County
  - Spitalul Clinic Sf. Maria /ID# 203809, Bucharest
  - Spitalul Clinic Colentina /ID# 204889, Bucharest
- Russia (6):
  - Kemerovo State Medical University /ID# 203676, Kemerovo, Kemerovo Oblast
  - Moscow Regional Research and Clinical Institute n.a. Vladimirskiy (MONIKI) /ID# 221643, Moscow, Moscow Oblast
  - Practicheskaya Medicina Clinic /ID# 224612, Moscow
  - First Moscow State Medical University n.a I.M. Sechenov /ID# 203673, Moscow
  - Euromedservice /ID# 205345, Pushkin
  - Clinical Rheumatologic Hospital No 25 /ID# 208950, Saint Petersburg
- Spain (10):
  - Complejo Hospitalario Universitario A Coruña /ID# 224731, A Coruña, A Coruna
  - Hospital Universitario Marques de Valdecilla /ID# 201604, Santander, Cantabria
  - Hospital Meixoeiro (CHUVI) /ID# 212084, Vigo, Pontevedra
  - Hospital Universitario Canarias /ID# 224928, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitario Basurto /ID# 224730, Bilbao, Vizcaya
  - Hospital Clinic de Barcelona /ID# 201878, Barcelona
  - Hospital Universitario Virgen de las Nieves /ID# 224726, Granada
  - Hospital General Universitario Gregorio Maranon /ID# 201326, Madrid
  - Hospital Clinico San Carlos /ID# 204871, Madrid
  - Hospital Universitario La Paz /ID# 241848, Madrid
- Sweden (6):
  - Skane University hospital /ID# 171407, Malmo, Skåne County
  - Karolinska University Hospital Solna /ID# 204945, Solna, Stockholm County
  - Uppsala University Hospital /ID# 171403, Uppsala, Uppsala County
  - Sahlgrenska Universitetssjukhuset /ID# 171405, Gothenburg, Västra Götaland County
  - Duplicate_Danderyds sjukhus /ID# 171404, Stockholm
  - Duplicate_Vastmanlands Sjukhus /ID# 171429, Västerås
- Switzerland (4):
  - Universitätsspital Basel /ID# 201767, Basel Town, Canton of Basel-City
  - Kantonsspital St. Gallen /ID# 201134, Sankt Gallen, Canton of St. Gallen
  - Inselspital, Universitaetsspital Bern /ID# 201364, Bern
  - HFR Fribourg - Hôpital cantonal /ID# 201114, Fribourg
- United Kingdom (9):
  - Royal United Hospitals Bath /ID# 239850, Bath, Bath And North East Somerset
  - Royal Devon & Exeter Hospital /ID# 202834, Exeter, Devon
  - University Hospitals Dorset NHS Foundation Trust /ID# 202836, Poole, Dorset
  - Barts Health NHS Trust /ID# 210511, London, Greater London
  - UH Coventry & Warwickshire /ID# 202838, Coventry, Warwickshire
  - Liverpool University University Hospitals NHS Foundation Trust /ID# 240391, Liverpool
  - Portsmouth Hospitals University NHS Trust /ID# 225002, Portsmouth
  - Southend Hospital /ID# 202839, Southend
  - Torbay and South Devon Nhs Foundation Trust /Id# 224689, Torquay

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Blockmans D, Penn SK, Setty AR, Schmidt WA, Rubbert-Roth A, Hauge EM, Keen HI, Ishii T, Khalidi N, Dejaco C, Cid MC, Hellmich B, Liu M, Zhao W, Lagunes I, Romero AB, Wung PK, Merkel PA; SELECT-GCA Study Group. A Phase 3 Trial of Upadacitinib for Giant-Cell Arteritis. N Engl J Med. 2025 May 29;392(20):2013-2024. doi: 10.1056/NEJMoa2413449. Epub 2025 Apr 2. PMID 40174237
- [Derived] Loricera J, Tofade T, Prieto-Pena D, Romero-Yuste S, de Miguel E, Riveros-Frutos A, Ferraz-Amaro I, Labrador E, Maiz O, Becerra E, Narvaez J, Galindez-Agirregoikoa E, Gonzalez-Fernandez I, Urruticoechea-Arana A, Ramos-Calvo A, Lopez-Gutierrez F, Castaneda S, Unizony S, Blanco R. Effectiveness of janus kinase inhibitors in relapsing giant cell arteritis in real-world clinical practice and review of the literature. Arthritis Res Ther. 2024 Jun 5;26(1):116. doi: 10.1186/s13075-024-03314-9. PMID 38840219
- See also: Description Related Info — https://www.abbvieclinicaltrials.com/study/?id=M16-852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 100 sites in 23 countries. Participants were randomized via in a 2:1:1 ratio to receive either upadacitinib 15 mg or 7.5 mg once daily in combination with a predefined 26-week CS taper regimen, or placebo with a predefined 52-week CS taper regimen
Pre-assignment Details: Those assigned to upadacitinib who achieved sustained remission for at least 24 consecutive weeks prior to Week 52 visit (at the end of Period 1) were re-randomized in a 2:1 ratio to either stay on upadacitinib or switch to placebo in Period 2. Those on placebo who achieved sustained remission for at least 24 weeks prior to Week 52 visit continued on placebo in Period 2.
Groups:
- Placebo + 52-week CS Taper: Participants randomized to receive placebo tablets for upadacitinib administered orally once daily (QD) for 52 weeks and a 52-week corticosteroid (CS) taper regimen during Period 1.
- 7.5 mg Upadacitinib + 26-week CS Taper: Participants randomized to receive 7.5 mg upadacitinib tablets administered orally once daily (QD) for 52 weeks and a 26-week corticosteroid (CS) taper regimen during Period 1.
- 15 mg Upadacitinib + 26-week CS Taper: Participants randomized to receive 15 mg upadacitinib tablets administered orally once daily (QD) for 52 weeks and a 26-week corticosteroid (CS) taper regimen during Period 1.
- Placebo + 52-week CS Taper -> Placebo: Participants who achieved sustained remission for at least 24 weeks prior to the Week 52 visit (at the end of Period 1) OR who had absence of GCA signs and symptoms and were CS-free at the Week 52 visit who were randomized to placebo tablets for upadacitinib administered orally once daily (QD) in Period 1 continued to receive placebo tablets for upadacitinib administered orally once daily (QD) in Period 2.
- 7.5 mg Upadacitinib + 26-week CS Taper -> 7.5 mg Upadacitinib: Participants randomized to receive 7.5 mg upadacitinib tablets administered orally once daily (QD) in Period 2.
- 7.5 mg Upadacitinib + 26-week CS Taper -> Placebo; 15 mg Upadacitinib + 26-week CS Taper -> Placebo: Participants randomized to receive placebo tablets for upadacitinib administered orally once daily (QD) in Period 2.
- 15 mg Upadacitinib + 26-week CS Taper -> 15 mg Upadacitinib: Participants randomized to receive 15 mg upadacitinib tablets administered orally once daily (QD) in Period 2.
Period: Period 1 (Baseline - Week 52)
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper | Placebo + 52-week CS Taper -> Placebo | 7.5 mg Upadacitinib + 26-week CS Taper -> 7.5 mg Upadacitinib | 7.5 mg Upadacitinib + 26-week CS Taper -> Placebo | 15 mg Upadacitinib + 26-week CS Taper -> 15 mg Upadacitinib | 15 mg Upadacitinib + 26-week CS Taper -> Placebo
Started | 112 | 107 | 210 | 0 | 0 | 0 | 0 | 0
Randomized | 112 | 107 | 210 | 0 | 0 | 0 | 0 | 0
Received Randomized Study Drug | 112 | 107 | 209 | 0 | 0 | 0 | 0 | 0
Completed | 86 | 85 | 177 | 0 | 0 | 0 | 0 | 0
Not Completed | 26 | 22 | 33 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 13 | 11 | 17 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrew consent | 5 | 6 | 10 | 0 | 0 | 0 | 0 | 0
Not completed — COVID-19 logistical restrictions | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Failure to meet continuation criteria | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other, not specified | 5 | 5 | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Did not receive randomized study drug | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (Week 52 - Week 104)
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper | Placebo + 52-week CS Taper -> Placebo | 7.5 mg Upadacitinib + 26-week CS Taper -> 7.5 mg Upadacitinib | 7.5 mg Upadacitinib + 26-week CS Taper -> Placebo | 15 mg Upadacitinib + 26-week CS Taper -> 15 mg Upadacitinib | 15 mg Upadacitinib + 26-week CS Taper -> Placebo
Started | 0 | 0 | 0 | 43 | 39 | 14 | 92 | 35
Completed | 0 | 0 | 0 | 20 | 27 | 9 | 58 | 22
Not Completed | 0 | 0 | 0 | 23 | 12 | 5 | 34 | 13
Not completed — Ongoing in Period 2 | 0 | 0 | 0 | 19 | 11 | 2 | 27 | 8
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 2
Not completed — Withdrew consent | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Failure to meet continuation criteria | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other, not specified | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set in Period 1 (FAS1): all randomized participants who received at least 1 dose of study drug in Period 1
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper | Total
Number analyzed (Participants) | 112 | 107 | 209 | 428
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (7.33) | 71.1 (7.55) | 70.8 (7.31) | 71.1 (7.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 80 | 156 | 313
  Male | 35 | 27 | 53 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 6 | 13
  Not Hispanic or Latino | 107 | 105 | 203 | 415
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 10 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 2 | 1 | 0 | 3
  White | 103 | 99 | 199 | 401
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Remission at Week 52
Description: Sustained remission is defined as having achieved absence of giant cell arteritis (GCA) signs and symptoms from Week 12 through Week 52, and adherence to the protocol-defined corticosteroid (CS) taper regimen.
Time Frame: From Week 12 to Week 52
Population: Full analysis set in Period 1 (FAS1): all randomized participants who received at least 1 dose of study drug in Period 1; non-responder imputation incorporating multiple imputation or non-responder imputation only if there were no missing data due to COVID-19 logistic restrictions was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper
Number analyzed (Participants) | 112 | 107 | 209
percentage of participants | 29.0 [20.6 to 37.5] | 41.1 [31.8 to 50.4] | 46.4 [39.6 to 53.2]
Statistical Analysis 1: Comparison: Placebo + 52-week CS Taper vs 15 mg Upadacitinib + 26-week CS Taper; 15 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — Across the strata, 95% CI for adjusted difference and p-value are calculated according to the Cochran-Mantel-Haenszel test adjusted for strata (Baseline CS dose (prednisone or prednisolone > 30 mg or ≤30 mg) and disease status (new onset or relapsing disease)) for the comparison of two treatment groups. Within each stratum, 95% CI for difference are calculated using normal approximation to the binomial distribution; p = 0.0019, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 17.1, 95% CI 2-sided [6.3 to 27.8] — Response rate difference = 15 mg Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo + 52-week CS Taper vs 7.5 mg Upadacitinib + 26-week CS Taper; 7.5 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0579, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 12.1, 95% CI 2-sided [-0.4 to 24.6] — Response rate difference = 7.5 mg Upadacitinib - Placebo

2. Secondary Outcome: Percentage of Participants Achieving Sustained Complete Remission From Week 12 Through Week 52
Description: Sustained complete remission is defined as having absence of giant cell arteritis (GCA) signs and symptoms from Week 12 through Week 52; normalization of erythrocyte sedimentation rate (ESR); normalization of high sensitivity C-reactive protein (hs-CRP) and adherence to the protocol-defined CS taper regimen.
Time Frame: Week 12 through Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper
Number analyzed (Participants) | 112 | 107 | 209
percentage of participants | 16.1 [9.3 to 22.9] | 26.2 [17.8 to 34.5] | 37.1 [30.5 to 43.7]
Statistical Analysis 1: Comparison: Placebo + 52-week CS Taper vs 15 mg Upadacitinib + 26-week CS Taper; 15 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 20.7, 95% CI 2-sided [11.3 to 30.2] — Response rate difference = 15 mg Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo + 52-week CS Taper vs 7.5 mg Upadacitinib + 26-week CS Taper; 7.5 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0699, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 9.9, 95% CI 2-sided [-0.8 to 20.6] — Response rate difference = 7.5 mg Upadacitinib - Placebo

3. Secondary Outcome: Cumulative Corticosteroid (CS) Exposure Through Week 52
Description: The cumulative exposure to corticosteroid(s) through Week 52 of the study was documented.
Time Frame: Baseline up to Week 52
Population: Full analysis set in Period 1 (FAS1): all randomized participants who received at least 1 dose of study drug in Period 1. As observed analysis; participants who did not have an evaluation on a scheduled visit were excluded from the analysis for that visit.
Measure: Median (95% Confidence Interval); unit: mg
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper
Number analyzed (Participants) | 90 | 86 | 180
mg | 2882.0 [2762.00 to 3253.00] | 1905.0 [1615.00 to 2265.00] | 1615.0 [1615.00 to 1635.00]
Statistical Analysis 1: Comparison: Placebo + 52-week CS Taper vs 15 mg Upadacitinib + 26-week CS Taper; 15 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — P-value is based on the van Elteren test, adjusting for the strata (Baseline CS dose (prednisone or prednisolone > 30 mg or ≤ 30 mg) and disease status (new onset or relapsing disease)); p < 0.0001, van Elteren test
Statistical Analysis 2: Comparison: Placebo + 52-week CS Taper vs 7.5 mg Upadacitinib + 26-week CS Taper; 7.5 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p < 0.0001, van Elteren test

4. Secondary Outcome: Time to First Disease Flare Through Week 52
Description: Disease flare is defined as an event determined by the investigator to represent recurrence of Giant Cell Arteritis (GCA) signs or symptoms or an erythrocyte sedimentation rate (ESR) measurement > 30 mm/hr (attributable to GCA) AND requiring an increase in corticosteroid (CS) dose.
Time Frame: Baseline up to Week 52
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper
Number analyzed (Participants) | 112 | 107 | 209
days | 323.0 [249.00 to NA] — Not calculable/estimable due to low number of participants with events | NA [316.00 to NA] — Not calculable/estimable due to low number of participants with events | NA [NA to NA] — Not calculable/estimable due to low number of participants with events
Statistical Analysis 1: Comparison: Placebo + 52-week CS Taper vs 15 mg Upadacitinib + 26-week CS Taper; 15 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — Treatment comparisons in the distribution of time-to-event between each upadacitinib group and the placebo are conducted using stratified log-rank test stratified by stratification factors (Baseline CS dose (prednisone or prednisolone > 30 mg or ≤ 30 mg) and disease status (new onset or relapsing disease). Within each stratum, 95% CI for difference are calculated using Cox proportional hazards model with stratification factors as covariates; p = 0.0025, Log-rank test; Cox Proportional Hazard = 0.57, 95% CI 2-sided [0.399 to 0.826]
Statistical Analysis 2: Comparison: Placebo + 52-week CS Taper vs 7.5 mg Upadacitinib + 26-week CS Taper; 7.5 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 4, analysis 1]; p = 0.1778, Log-rank test; Cox Proportional Hazard = 0.75, 95% CI 2-sided [0.499 to 1.136]

5. Secondary Outcome: Percentage of Participants Who Experience at Least 1 Disease Flare Through Week 52
Description: The percentage of participants who experience at least 1 disease flare was calculated. Disease flare is defined as an event determined by the investigator to represent recurrence of Giant Cell Arteritis (GCA) signs or symptoms or an erythrocyte sedimentation rate (ESR) measurement > 30 mm/hr (attributable to GCA) AND requiring an increase in corticosteroid (CS) dose.
Time Frame: Baseline up to Week 52
Population: Full analysis set in Period 1 (FAS1): all randomized participants who received at least 1 dose of study drug in Period 1; as observed analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper
Number analyzed (Participants) | 112 | 107 | 209
percentage of participants | 55.6 [42.9 to 69.2] | 41.3 [32.2 to 51.7] | 34.3 [27.4 to 42.4]
Statistical Analysis 1: Comparison: Placebo + 52-week CS Taper vs 15 mg Upadacitinib + 26-week CS Taper; 15 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — The point estimate of flare rate at Week 52 from the Kaplan-Meier estimate for each stratum is used to derive the stratified disease flare rate. P-value, and 95% CI for the odds ratio between each upadacitinib group and placebo is also provided. Stratification factors (Baseline CS dose (prednisone or prednisolone > 30 mg or ≤ 30 mg) and disease status (new onset or relapsing disease) were used; p = 0.0014, Stratified Test for Odds Ratio; This method is described in J Immunother Cancer. 2021 Nov;9(11):e003323. doi: 10.1136/jitc-2021-003323; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.29 to 0.74]
Statistical Analysis 2: Comparison: Placebo + 52-week CS Taper vs 7.5 mg Upadacitinib + 26-week CS Taper; 7.5 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.0633, Stratified Test for Odds Ratio; This method is described in J Immunother Cancer. 2021 Nov;9(11):e003323. doi: 10.1136/jitc-2021-003323; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.35 to 1.03]

6. Secondary Outcome: Percentage of Participants in Complete Remission at Week 52
Description: Complete remission is defined as having achieved absence of Giant Cell Arteritis (GCA) signs and symptoms; normalization of erythrocyte sedimentation rate (ESR) to < 30 mm/hr-- if ESR ≥30 mm/hr and elevation is not attributable to GCA, this criterion can still be met); normalization of high sensitivity C-reactive protein (hs-CRP) to < 1 mg/dL; and adherence to the protocol-defined corticosteroid (CS) taper regimen.
Time Frame: At Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper
Number analyzed (Participants) | 112 | 107 | 209
percentage of participants | 19.6 [12.3 to 27.0] | 43.0 [33.6 to 52.4] | 50.2 [43.4 to 57.1]
Statistical Analysis 1: Comparison: Placebo + 52-week CS Taper vs 15 mg Upadacitinib + 26-week CS Taper; 15 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 30.3, 95% CI 2-sided [20.4 to 40.2]
Statistical Analysis 2: Comparison: Placebo + 52-week CS Taper vs 7.5 mg Upadacitinib + 26-week CS Taper; 7.5 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 23.5, 95% CI 2-sided [11.7 to 35.3]

7. Secondary Outcome: Percentage of Participants in Complete Remission at Week 24
Description: as for outcome 6
Time Frame: At Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper
Number analyzed (Participants) | 112 | 107 | 209
percentage of participants | 36.1 [27.2 to 45.1] | 39.3 [30.0 to 48.5] | 57.2 [50.5 to 64.0]
Statistical Analysis 1: Comparison: Placebo + 52-week CS Taper vs 15 mg Upadacitinib + 26-week CS Taper; 15 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0002, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 20.8, 95% CI 2-sided [9.7 to 31.9]
Statistical Analysis 2: Comparison: Placebo + 52-week CS Taper vs 7.5 mg Upadacitinib + 26-week CS Taper; 7.5 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.6276, Cochran-Mantel-Haenszel; Adjusted Response Rate Difference = 3.2, 95% CI 2-sided [-9.6 to 16.0]

8. Secondary Outcome: Change From Baseline in the 36-item Short Form Quality of Life Questionnaire (SF-36) Physical Component Summary (PCS) Score at Week 52
Description: The Short Form 36-Item Health Survey (SF-36) Version 2 is a self-administered questionnaire that measures the impact of disease on overall quality of life during the past 4 weeks. The SF-36 consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health).
  The physical component summary (PCS) is a weighted combination of the 8 subscales with positive weighting for physical functioning, role-physical, bodily pain, and general health. The SF-36 PCS ranges from 0 to 100. A linear algorithm was applied to the calculation of the PCS which has a normative mean value of 50. Higher scores are associated with less disability; a score of 100 is equivalent to no disability and a score of 0 is equivalent to maximum disability. A positive change from the Baseline score indicates improvement.
Time Frame: Baseline, Week 52
Population: Full analysis set in Period 1 (FAS1): all randomized participants who received at least 1 dose of study drug in Period 1 with both Baseline and post-Baseline visit values
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper
Number analyzed (Participants) | 44 | 49 | 123
units on a scale | -1.2892 [-3.3093 to 0.7309] | 1.3202 [-0.6553 to 3.2957] | 2.4634 [1.1707 to 3.7561]
Statistical Analysis 1: Comparison: Placebo + 52-week CS Taper vs 15 mg Upadacitinib + 26-week CS Taper; 15 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — The Mixed-Effect Model Repeat Measurement with Baseline value, categorical fixed effects of treatment, visit and treatment-by-visit interaction, stratification factors at randomization (Baseline CS dose (prednisone or prednisolone >30 mg, prednisone or prednisolone ≤30 mg) and Baseline disease status (new onset disease, relapsing disease)) included in the model. An unstructured variance covariance matrix is used. Data after initiation of corticosteroid escape therapy are excluded from the model; p = 0.0019, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 3.7526, 95% CI 2-sided [1.3932 to 6.1119], Standard Error of Mean 1.1981 — Difference = 15 mg Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo + 52-week CS Taper vs 7.5 mg Upadacitinib + 26-week CS Taper; 7.5 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0670, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 2.6094, 95% CI 2-sided [-0.1841 to 5.4028], Standard Error of Mean 1.4185 — Difference = 7.5 mg Upadacitinib - Placebo

9. Secondary Outcome: Number of Disease Flares Per Participant Through Week 52
Description: The number of disease flares per participant during Period 1 was documented, and was adjusted by the duration of study participation.
Time Frame: Baseline up to Week 52
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Disease Flare per Participant per Year
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper
Number analyzed (Participants) | 112 | 107 | 209
Disease Flare per Participant per Year | 0.7 [0.5 to 0.9] | 0.6 [0.4 to 0.7] | 0.4 [0.3 to 0.5]
Statistical Analysis 1: Comparison: Placebo + 52-week CS Taper vs 15 mg Upadacitinib + 26-week CS Taper; 15 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — Comparisons between each upadacitinib treatment group and the placebo group are carried out using Poisson regression model with stratification factors as covariates and log(duration of study participation in years) as an offset. Robust standard error is used in inference; p = 0.0010, Poisson regression model; Rate Ratio = 0.6, 95% CI 2-sided [0.4 to 0.8]
Statistical Analysis 2: Comparison: Placebo + 52-week CS Taper vs 7.5 mg Upadacitinib + 26-week CS Taper; 7.5 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.2722, Poisson regression model; Rate Ratio = 0.8, 95% CI 2-sided [0.6 to 1.2]

10. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) at Week 52
Description: The FACIT-Fatigue questionnaire is a self-administered patient questionnaire that consists of 13 questions designed to measure the degree of fatigue experienced by participants in the previous 7 days, including physical fatigue, functional fatigue, emotional fatigue, and social consequences of fatigue. Participants respond to the questions on a scale from 0 (not at all) to 4 (very much). The FACIT-Fatigue score is computed by summing the item scores, after reversing items worded in the negative direction. The FACIT-Fatigue score ranges from 0 to 52, where higher scores represent less fatigue. A positive change from Baseline indicates improvement.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper
Number analyzed (Participants) | 45 | 49 | 123
units on a scale | -2.4 [-4.71 to -0.07] | 1.1 [-1.17 to 3.37] | 1.7 [0.18 to 3.14]
Statistical Analysis 1: Comparison: Placebo + 52-week CS Taper vs 15 mg Upadacitinib + 26-week CS Taper; 15 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0036, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 4.0, 95% CI 2-sided [1.33 to 6.76], Standard Error of Mean 1.38 — Difference = 15 mg Upadacitinib -Placebo
Statistical Analysis 2: Comparison: Placebo + 52-week CS Taper vs 7.5 mg Upadacitinib + 26-week CS Taper; 7.5 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.0338, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 3.5, 95% CI 2-sided [0.27 to 6.70], Standard Error of Mean 1.63 — Difference = 7.5 mg Upadacitinib -Placebo

11. Secondary Outcome: Assessment of Treatment Satisfaction Questionnaire for Medication (TSQM) Patient Global Satisfaction Subscale at Week 52
Description: The Treatment Satisfaction Questionnaire for Medications (TSQM) is a generic ePRO measure of treatment satisfaction, developed to compare treatment satisfaction between medication types and conditions. TSQM comprises of 14 items to assess 4 domains (effectiveness, side effects, convenience, and global satisfaction). The TSQM items are rated on a Likert scale (1 = extremely dissatisfied to 7 = extremely satisfied). Scores for each of the 4 domains range from 0 to 100, with higher scores corresponding to higher satisfaction. A positive change from Baseline indicates improvement.
Time Frame: At Week 52
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper
Number analyzed (Participants) | 45 | 52 | 126
units on a scale | 68.8428 [63.8310 to 73.8547] | 74.2644 [69.4483 to 79.0805] | 71.5753 [68.3375 to 74.8131]
Statistical Analysis 1: Comparison: Placebo + 52-week CS Taper vs 15 mg Upadacitinib + 26-week CS Taper; 15 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.3573, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 2.7325, 95% CI 2-sided [-3.1020 to 8.5670], Standard Error of Mean 2.9635 — Difference = 15 mg Upadacitinib -Placebo
Statistical Analysis 2: Comparison: Placebo + 52-week CS Taper vs 7.5 mg Upadacitinib + 26-week CS Taper; 7.5 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.1203, Mixed-Effect Model Repeat Measurement; LS Mean Difference = 5.4216, 95% CI 2-sided [-1.4269 to 12.2701], Standard Error of Mean 3.4785 — Difference = 7.5 mg Upadacitinib -Placebo

12. Secondary Outcome: Rate of Corticosteroid-related Adverse Events Though Week 52
Description: The rate of corticosteroid-related adverse events was calculated, and was adjusted by duration of study drug exposure.
Time Frame: Baseline up to Week 52
Population: Safety Analysis Set in Period 1: all participants who received at least 1 dose of study drug in Period 1
Measure: Mean (95% Confidence Interval); unit: CS-related AE per participant per year
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper
Number analyzed (Participants) | 112 | 107 | 209
CS-related AE per participant per year | 1.7 [1.3 to 2.3] | 1.7 [1.2 to 2.2] | 2.0 [1.7 to 2.4]
Statistical Analysis 1: Comparison: Placebo + 52-week CS Taper vs 15 mg Upadacitinib + 26-week CS Taper; 15 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.4371, Poisson regression model; Rate Ratio = 1.1, 95% CI 2-sided [0.8 to 1.6]
Statistical Analysis 2: Comparison: Placebo + 52-week CS Taper vs 7.5 mg Upadacitinib + 26-week CS Taper; 7.5 mg Upadacitinib + 26-week CS taper vs Placebo + 52-week CS taper; Test type: Superiority — [test comment as in outcome 9, analysis 1]; p = 0.7749, Poisson regression model; Rate Ratio = 0.9, 95% CI 2-sided [0.6 to 1.4]

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse events were collected from the time informed consent was signed through 06 February 2024. Median time on follow-up was for 378 days for Pbo (Period 1); 377 days for Upa 7.5 mg (Period 1); 378 days for Upa 15 mg (Period 1); 289 days for Pbo -> Pbo (Period 2); 364 days for 7.5 mg Upa -> 7.5 mg Upa (Period 2); 348 days for 7.5 mg Upa -> Pbo (Period 2); 363.5 days for 15 mg Upa -> 15 mg Upa (Period 2); and 363 days for 15 mg Upa -> Pbo (Period 2).
Groups:
- 15 mg Upadacitinib + 26-week CS Taper -> 15 mg Upadacitinib: Participants randomized to receive15 mg upadacitinib tablets administered orally once daily (QD) in Period 2.
Arm/Group | Placebo + 52-week CS Taper | 7.5 mg Upadacitinib + 26-week CS Taper | 15 mg Upadacitinib + 26-week CS Taper | Placebo + 52-week CS Taper -> Placebo | 7.5 mg Upadacitinib + 26-week CS Taper -> 7.5 mg Upadacitinib | 7.5 mg Upadacitinib + 26-week CS Taper -> Placebo | 15 mg Upadacitinib + 26-week CS Taper -> 15 mg Upadacitinib | 15 mg Upadacitinib + 26-week CS Taper -> Placebo
All-Cause Mortality (participants affected / at risk) | 2/112 | 0/107 | 3/210 | 0/43 | 0/39 | 0/14 | 0/92 | 0/35
Serious Adverse Events (participants affected / at risk) | 24/112 | 14/107 | 50/210 | 6/43 | 5/39 | 0/14 | 11/92 | 4/35
Other Adverse Events (participants affected / at risk) | 88/112 | 88/107 | 174/210 | 27/43 | 21/39 | 12/14 | 61/92 | 30/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + 52-week CS Taper (N=112) | 7.5 mg Upadacitinib + 26-week CS Taper (N=107) | 15 mg Upadacitinib + 26-week CS Taper (N=210) | Placebo + 52-week CS Taper -> Placebo (N=43) | 7.5 mg Upadacitinib + 26-week CS Taper -> 7.5 mg Upadacitinib (N=39) | 7.5 mg Upadacitinib + 26-week CS Taper -> Placebo (N=14) | 15 mg Upadacitinib + 26-week CS Taper -> 15 mg Upadacitinib (N=92) | 15 mg Upadacitinib + 26-week CS Taper -> Placebo (N=35)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENDOCARDITIS FIBROPLASTICA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOXIC NODULAR GOITRE (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIPLOPIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GLAUCOMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MACULAR OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROINTESTINAL ANGIODYSPLASIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEATH (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPERGILLUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ERYSIPELAS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEBRILE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS CLOSTRIDIAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENITOURINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISCITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PNEUMONIA BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SALMONELLOSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEPTIC ARTHRITIS STREPTOCOCCAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UROSEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TROPONIN T INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MENISCAL DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VERTEBRAL FORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT NEOPLASM OF AMPULLA OF VATER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYXOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROSTATIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TONSIL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBELLAR ATAXIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL AMYLOID ANGIOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBROSPINAL FISTULA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
QUADRANTANOPIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBSTANCE-INDUCED PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AORTIC DISSECTION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AORTIC THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTERIOSCLEROSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GIANT CELL ARTERITIS (Vascular disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL EMBOLISM (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + 52-week CS Taper (N=112) | 7.5 mg Upadacitinib + 26-week CS Taper (N=107) | 15 mg Upadacitinib + 26-week CS Taper (N=210) | Placebo + 52-week CS Taper -> Placebo (N=43) | 7.5 mg Upadacitinib + 26-week CS Taper -> 7.5 mg Upadacitinib (N=39) | 7.5 mg Upadacitinib + 26-week CS Taper -> Placebo (N=14) | 15 mg Upadacitinib + 26-week CS Taper -> 15 mg Upadacitinib (N=92) | 15 mg Upadacitinib + 26-week CS Taper -> Placebo (N=35)
CATARACT (Eye disorders) | 2 (2) | 6 (7) | 10 (10) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
OCULAR HYPERAEMIA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 (5) | 0 (0) | 11 (13) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 8 (8) | 11 (11) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 12 (12) | 5 (6) | 17 (20) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 4 (6) | 6 (7) | 11 (17) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 6 (6) | 4 (4) | 18 (21) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
MALAISE (General disorders) | 1 (1) | 0 (0) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OEDEMA PERIPHERAL (General disorders) | 2 (3) | 7 (8) | 15 (16) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
PERIPHERAL SWELLING (General disorders) | 3 (3) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 8 (9) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 12 (12) | 12 (12) | 27 (28) | 7 (7) | 6 (6) | 3 (3) | 15 (15) | 6 (6)
CYSTITIS (Infections and infestations) | 3 (3) | 5 (5) | 14 (19) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 13 (14) | 6 (7) | 18 (21) | 2 (2) | 4 (5) | 0 (0) | 6 (6) | 3 (4)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (2)
SINUSITIS (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
TOOTH INFECTION (Infections and infestations) | 3 (3) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (10) | 8 (8) | 11 (11) | 2 (2) | 0 (0) | 2 (3) | 4 (4) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 17 (26) | 15 (18) | 21 (25) | 1 (3) | 3 (3) | 1 (1) | 4 (4) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 7 (8) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 4 (4) | 4 (6) | 7 (7) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GLUCOSE URINE PRESENT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OCCULT BLOOD POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
WEIGHT INCREASED (Investigations) | 4 (4) | 6 (6) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 15 (16) | 7 (8) | 29 (33) | 8 (8) | 0 (0) | 1 (1) | 10 (10) | 3 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 14 (15) | 6 (7) | 25 (28) | 1 (1) | 0 (0) | 1 (1) | 5 (5) | 3 (3)
GREATER TROCHANTERIC PAIN SYNDROME (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6) | 13 (13) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (9) | 9 (9) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 11 (12) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4) | 15 (16) | 2 (2) | 0 (0) | 0 (0) | 6 (7) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
DIZZINESS (Nervous system disorders) | 6 (6) | 6 (7) | 10 (10) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
HEADACHE (Nervous system disorders) | 13 (14) | 16 (23) | 33 (46) | 1 (2) | 3 (3) | 0 (0) | 11 (12) | 1 (2)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (8) | 14 (16) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 11 (11) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GIANT CELL ARTERITIS (Vascular disorders) | 34 (41) | 27 (34) | 45 (57) | 7 (9) | 2 (2) | 4 (4) | 8 (8) | 13 (18)
HYPERTENSION (Vascular disorders) | 13 (13) | 16 (17) | 28 (31) | 1 (1) | 1 (1) | 0 (0) | 5 (6) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/02/NCT03725202/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT03725202/SAP_001.pdf